CLINICAL TRIAL: NCT06260176
Title: A Large Scale Long-term Randomized Trial of Nutrition Labeling Interventions
Brief Title: Vending Labeling Sales and Intercepts Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 828722; R01DK113307 (NIH); 15163 (Registry Identifier: AsPredicted.org)
Record Dates: First submitted 2024-01-29; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Food Preferences; Obesity; Weight Gain
Keywords: food labeling; sugar-sweetened beverages; eating; drinking; choice behavior
MeSH Terms: conditions — Food Preferences; Obesity; Weight Gain

STUDY DESIGN:
Intervention Model Description: Machine locations were randomly assigned to 1 of 4 front-of-package message arms, stratified by baseline machine sales (high/low) and type of machine location (correctional facilities, courts/offices, large offices, police/fire, recreation centers/libraries/other) with equal probability. The investigators first randomized vending locations (e.g., floors) with beverage machines so that all machines on the same floor displayed the same label. They then randomized the remaining "solo" snack locations. Monthly sales data provided by the City's vending contractor indicated consumer choices. Research assistants also asked a subset of consumers (N=1,065) about their purchases. Intercepts were not allowed in the courts/offices location type and were not conducted at correctional facilities with low traffic. The aim was to collect 10 intercepts per machine visited, distributed over the entire study period, however the study was cut short in March 2020 by the Covid pandemic.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Green labels (Experimental): green label added to healthy product slots; no additional labels shown for "less healthy" products and 1 poster per machine explaining the labels
  Interventions: Behavioral: exposure to healthy labels only
- Traffic light labels (Experimental): red/yellow/green labels added to slots for less healthy/moderately healthy/healthy products, respectively and 1 poster per machine explaining the labels
  Interventions: Behavioral: exposure to healthiness information
- Physical activity calorie equivalent labels (Experimental): labels added to slots that display products' calorie content in terms of physical activity required to burn those calories and 1 poster per machine explaining the labels
  Interventions: Behavioral: exposure to physical activity equivalents
- Sweetened beverage tax posters (Experimental): 1 poster per machine; no labels; posters reminded consumers of the Philadelphia sweetened beverage tax and encouraging healthier choices
  Interventions: Behavioral: exposure to sweetened beverage tax messaging

INTERVENTIONS:
Behavioral: exposure to healthy labels only — Green labels only for beverages and foods scored as healthy
  Arms: Green labels
Behavioral: exposure to healthiness information — All beverages and foods labeled as either healthy (green), moderately healthy (yellow), or less healthy (red)
  Arms: Traffic light labels
Behavioral: exposure to physical activity equivalents — All beverages and foods labeled with physical activity required to burn their calories
  Arms: Physical activity calorie equivalent labels
Behavioral: exposure to sweetened beverage tax messaging — Message reminding consumers to make healthier choices
  Arms: Sweetened beverage tax posters

SUMMARY:
The aim of this study is to compare the impact of 4 different types of front of package (FOP) food and beverage messages: 1) green labels on healthy foods, 2) red/yellow/green labels on less healthy/moderately healthy/healthy foods, 3) physical activity calorie equivalent labels, and 4) posters reminding consumers of the sweetened beverage tax on consumers' beverage and snack selections.

DETAILED DESCRIPTION:
This project involves a randomized field experiment. The investigators worked with the vending contractor for the City of Philadelphia to randomize vending machine locations (covering ~260 beverage and snack machines) to one of the four different message conditions: 1) single green traffic light labels (on healthy foods); 2) multiple traffic light labels (red traffic light labels applied to less healthy foods, yellow applied to moderately healthy foods, and green on healthy foods); 3) physical activity labels (calorie content displayed in terms of physical activity equivalents); 4) posters reminding consumers of the Philadelphia sweetened beverage tax and encouraging healthier choices. The City's vending machine contractors provided monthly aggregated sales data from each machine for analysis. Customer intercepts were also collected at the point of sale, after customers completed their purchase, to evaluate factors that moderate message influence. They were asked to answer questions about their perceptions of the different labels.

ELIGIBILITY:
Sales data include all purchases at the machine regardless of customer demographics.

Customer purchase assessment data were collected from:

Inclusion Criteria:

* Any person aged 18 or older making a purchase from the vending machines included in this intervention will be asked to participate in this study.

Exclusion Criteria:

* People who indicate they have already taken the survey are not eligible to take the survey again.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1065 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Percentage of beverages sold with calories per month | Every month, for 13 months
  Outcome is percentage of monthly beverages selected that had calories
Calories sold from beverages per month, if beverages with calories sold | Every month, for 13 months
  Outcome is calories in beverages sold per month - only for beverages with calories.
Calories sold from snacks per month | Every month, for 13 months
  Outcome is calories in snacks sold per month.
Likelihood of selecting a healthy beverage | Every month, for 13 months
  Outcome is percentage of monthly beverages selected were healthy beverages (green labeled in the traffic light condition)
Likelihood of selecting a moderately healthy beverage | Every month, for 13 months
  Outcome is percentage of monthly beverages selected were moderately healthy beverages (yellow labeled in the traffic light condition)
Likelihood of selecting a less healthy beverage | Every month, for 13 months
  Outcome is percentage of monthly beverages selected were less healthy beverages (red labeled in the traffic light condition)
Likelihood of selecting a healthy snack | Every month, for 13 months
  Outcome is percentage of monthly snacks selected were healthy snacks (green labeled in the traffic light condition)
Likelihood of selecting a moderately healthy snack | Every month, for 13 months
  Outcome is percentage of monthly snacks selected were moderately healthy snacks (yellow labeled in the traffic light condition)
Likelihood of selecting a less healthy snack | Every month, for 13 months
  Outcome is percentage of monthly snacks selected were less healthy snacks (red labeled in the traffic light condition)
Total beverage units sold per month per machine. | Every month, for 13 months
  Outcome is number of monthly beverages sold per machine
Total snack units sold per month per machine | Every month, for 13 months
  Outcome is number of monthly snacks sold per machine

SECONDARY OUTCOMES:
Total revenue per month per beverage machine | Every month, for 13 months
  Outcome is the total dollar sales per month per beverage machine.
Total revenue per month per snack machine | Every month, for 13 months
  Outcome is the total dollar sales per month per snack machine.
Total calories sold per customer trip | 5-minute survey
  Customer purchase assessments will be conducted in front of study machines. Outcome is total number of calories (beverage + snack) purchased per customer trip.

CONTACTS AND LOCATIONS:
Overall Officials: Christina A Roberto, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Machine sales data are proprietary and cannot be shared. However, no identifiable data were collected from the customer purchase assessments, so after analysis, the investigators will upload the customer de-identified data to ResearchBox for public sharing.
Supporting Information: SAP
Time Frame: starting 6 months after publication
Access Criteria: public

REFERENCES:
- [Derived] Gibson LA, Stephens-Shields AJ, Hua SV, Orr JA, Lawman HG, Bleich SN, Volpp KG, Bleakley A, Thorndike AN, Roberto CA. Comparison of Sales From Vending Machines With 4 Different Food and Beverage Messages: A Randomized Trial. JAMA Netw Open. 2024 May 1;7(5):e249438. doi: 10.1001/jamanetworkopen.2024.9438. PMID 38717775